CLINICAL TRIAL: NCT03600961
Title: BIOTRONIK - SaFety and Performance Registry for an Allcomers Patient Population With the SiroLimus Eluting Orsiro Stent Within Daily Clinical Practice in Small Vessels - Portugal Registry
Brief Title: BIOFLOW-SV Portugal Registry
Acronym: BIOFLOW-SV
Status: Terminated | Type: Observational
Why Stopped: Problem with enrollment due to Covid-19
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Other Study IDs: C1704
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Orsiro Sirolimus Eluting Coronary Stent System — Percutaneous coronary intervention

SUMMARY:
Assessment of the clinical safety and performance of the Orsiro drug-eluting stent in a real world setting in patients with small vessels with reference vessel diameter ≤2.75 mm

DETAILED DESCRIPTION:
Prospective, single-arm, multi-center, all-comers registry with clinical follow-up visits at the hospital or by phone at 6 and 12 months post-procedure. A minimum of 1000 patients will be enrolled in approximately 15 sites in Brazil, including at least 415 patients with reference vessel diameter ≤2.75 mm as assessed by online QCA.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years of age
* Subject must sign a Patient Informed Consent (PIC) or a Patient Data Release Form (PDRF)
* Subject must agree to undergo all required follow-up visits

Exclusion Criteria:

* Pregnant and/or breast feeding females at the time of enrolment
* Known allergies to Acetylsalicylic Acid (ASA), clopidogrel, ticlopidin, heparin or any other anticoagulant

  /antiplatelet required for PCI, contrast medium, sirolimus, or similar drugs, or the stent materials that cannot be adequately pre-medicated
* Currently participating in another study that has not yet reached the primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This registry will include subjects requiring a treatment of coronary artery disease with an Orsiro DES
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Target Lesion Failure for the small vessel group | at 12 months
  Primary endpoint will be Target Lesion Failure (TLF) at 12 months for the small vessels group, defined as a composite of cardiac death, target vessel Myocardial Infarction (MI) or clinically driven Target Lesion Revascularization (TLR)

SECONDARY OUTCOMES:
TLF for the overall cohort | at 12 months
  TLF at 12 months post procedure for the overall cohort
Clinically driven Target Lesion Revascularization (TLR) | at 6 and 12 months
  Clinically driven Target Lesion Revascularization (TLR) at 6 and 12 months post procedure
Clinically driven Target Vessel Revascularization (TVR) | at 6 and 12 months
  Clinically driven Target Vessel Revascularization (TVR) at 6 and 12 months post procedure
Definite and probable stent thrombosis | at 6 and 12 months
  Definite and probable stent thrombosis at 6 and 12 months post procedure (ARC Definition)
Procedure success | 12 months
  defined as achievement of a final diameter stenosis of <30% by investigator's visual estimate (using any percutaneous method) without the occurrence of death, MI, or repeat revascularization of the target lesion during the hospital stay
Device success | 12 months
  defined as a final residual diameter stenosis of <30% by investigator's visual estimate, using the assigned device only, successful delivery of the stent to the target lesion site in the coronary artery, appropriate stent deployment, and successful removal of the device. Post-dilatation is allowed to achieve device success

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Braga, MD, Principal Investigator — Centro Hospitalar de Vila Nova de Gaia
Locations (4):
- Portugal (4):
  - Hospital de Santa Cruz, Carnaxide
  - Hospital da Luz, Carnaxide
  - Hospital Espirito Santo Evora, Evora
  - Centro Hospitaler de Leiria E.P.E., Leiria

IPD SHARING:
Plan to Share IPD: No